CLINICAL TRIAL: NCT06314035
Title: "Effects of a Decision Support Intervention on End-of-life Care Planning in Chinese Older Adults With Advanced Disease and Their Family Members: A Feasibility Trial"
Brief Title: Decision Support on End-of-life Care Planning in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai Ching Ting, Jenny, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIC2023003
Record Dates: First submitted 2024-03-03; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; advance care planning; decision aid; readiness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to their group assignment. The personnel administering the interventions will not be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in experimental group will receive a COPD Decision Support Tool (PDA intervention).
  Interventions: Other: COPD Patient Decision Aid
- Attention Control Placebo Group (Placebo Comparator): Participants in the attention control placebo group will receive a general health coaching intervention. Dose and time similar to experimental group.
  Interventions: Other: General Health Coaching Intervention

INTERVENTIONS:
Other: COPD Patient Decision Aid — Participants in this group will receive two 60-minute intervention sessions in one month. The COPD PDA consists of three main parts: The first component, clinical counselling, guides the participants in reviewing the common EOL scenarios. The second component, an evidence-based decision aid, is presented as an option grid in a booklet and a video to provide information about outcome probabilities of various treatment options and survival estimates in a balanced and unbiased manner. The information is presented in plain language for laypersons. The third component, decision coaching, introduces the concept of ACP and guides deliberation through value clarification.
  Other Names: Experimental Group
  Arms: Experimental Group
Other: General Health Coaching Intervention — The participants in the control group will receive two 60-minute health coaching sessions developed by the PI for another project as an attention placebo control. Trained research personnel will use the same amount of interaction time and similar formats to avoid threats to the study's internal validity. This intervention will focus on lifestyle modification and self-care management unrelated to the tested intervention content or outcomes. The trained research personnel will give the guidebook consisting of general self-management advice to participants in this group.
  Other Names: Attention Control Placebo Group
  Arms: Attention Control Placebo Group

SUMMARY:
This study aims to test the effects of a patient decision aid (PDA) on planning for end-of-life (EOL) care among older adults with COPD. The main questions it aims to answer are:

1. Does a PDA improve the process of a person to make decisions on EOL care?
2. Does a PDA improve the readiness of a person to join advance care planning (ACP) communication?
3. Does a person make an advance directive after using a PDA?

Participants in this study will:

1. Be randomly assigned to one of two groups.
2. In the experimental group, participants will receive two 60-minute interactive consultations over four weeks, using a PDA to help clarify values and preferences for future medical care. A guidebook summarising these future care options will be provided.
3. In the control group, participants will receive two 60-minute sessions on lifestyle modification and self-care management over four weeks using a guidebook with coaching. A guidebook summarising general health information will be provided.

Researchers will compare the intervention group to the control group to see if the PDA is better at improving the decision-making process on EOL care, the readiness of a person to join ACP communication and the chance to make an advance directive.

DETAILED DESCRIPTION:
I. Research Background:

Chronic Obstructive Pulmonary Disease (COPD) is a progressive life-limiting condition and one of the leading causes of death globally and locally(MacPherson et al., 2013). Patients with COPD experience increasing symptom burden as the disease progresses, resulting in repeated episodes of exacerbation and hospital admissions(Sapey & Stockley, 2006). However, they and their family members are generally unprepared for the health changes and the perceived "sudden" changes often lead to care incongruent with patients' preferences, compromised quality of life and mistrust towards the healthcare team. Despite the projected disease progression, interventions or mechanisms to discuss end-of-life (EOL) care have not been systematically introduced in the management of COPD (Momen et al., 2012).

Advance care planning (ACP) aims to support people to plan for EOL and communicate their care wishes with family and the healthcare team before they lose mental capacity (Rietjens et al., 2017). ACP is gaining increased attention from the public. However, studies have shown that patients and their family members were unprepared for ACP due to unrealistic expectations towards medical treatments and cultural taboos of discussing death-related issues(Chan et al., 2018; Cheng et al., 2019). Conventional ACP interventions have positive but limited effects on empowering patients or EOL care decision-making. Studies reporting the effects of ACP on patients' readiness, decisional conflict, and the concordance between care preferences and the EOL care provided are mixed (Bravo et al., 2016; Cohen et al., 2019; Michael et al., 2022).

Decision aids have been developed as tools to support patients in making informed and preference-sensitive treatment decisions, with some explicitly for ACP(Cardona-Morrell et al., 2017; Elwyn et al., 2006). A Cochrane review found that decision aids are effective in reducing decisional conflict, clarifying personal values, increasing decision-making behaviours and improving patient-doctor communication(Stacey et al., 2017). However, the effects of a locally-adapted disease-specific decision aid for COPD, on decision-making are lacking.

II. Research Objectives:

This study aims to assess the effectiveness of PDA in improving the understanding of ACP and EOL medical care among individuals diagnosed with Chronic COPD. The specific research objectives are as follows:

1. Assess the practicality of implementing PDAs for individuals with COPD.
2. Evaluate the thoroughness with which PDA address the needs of COPD patients.
3. Determine COPD patients' acceptance of PDA.
4. Assess the practicality of the research measurement tools.
5. Evaluate the effectiveness of strategies for recruiting participants.
6. Examine participant completion rates and analyse dropout causes.
7. Explore the experiences of participants using the PDA.

III. Research Methodology:

(I) Research Design:

This 12-month study adopts a mixed-methods approach, incorporating the following procedures:

1. Quantitative Survey: We will conduct a single-blinded, randomised controlled trial (RCT) to assess the intervention's efficacy and impact systematically.
2. Qualitative Interviews: Semi-structured interviews will gather detailed insights into participants' experiences and perceptions regarding ACP, EOL treatment, and their interactions with the PDA.

(II) Study Population, Location, and Sample Size:

1. Location: The study targets individuals diagnosed with Chronic Obstructive Pulmonary Disease (COPD) in the northern community of Taiwan. Recruitment will occur across various settings, including community care points, nursing homes, and neighbourhood activity centres.
2. Sample Size: We have determined the required sample size for this study based on prior research conducted by our team on severe disease patients and their families concerning ACP in community settings (Chan et al., 2018). The primary objective is to evaluate decisional conflicts regarding EOL care, measured through SURE test scores, with effect sizes (Cohen's d) of 0.26 and 0.47 at one and six months, respectively (Chan et al., 2018). Factoring in a 35% dropout rate, as observed in our previous ACP studies (Bell et al., 2018; Chan et al., 2018; Julious, 2005), and using the empirical rule, the study necessitates 120 participants, equating to 60 individuals per group.
3. Subject Recruitment: The research team will partner with community care points, nursing homes, and neighbourhood activity centres in the northern region of Taiwan. The Principal Investigator (PI) will obtain approval from the leaders of these facilities to conduct the study and to place recruitment posters. Social workers or nurses at these community centres will initially screen for eligibility and manage the registration process.

(III) Informed consent, randomisation and blinding:

1. Informed Consent: Trained research personnel will evaluate participants' eligibility according to the inclusion criteria. Before any intervention, the research team will explain the informed consent form to the participants, ensuring they fully understand its contents. Following this, the team will ask participants to sign the consent form.
2. Randomisation and Blinding: This study will adopt a single-blind, random allocation approach. Before the commencement of the research activities, a computer-generated randomisation process will allocate participants to either the experimental or control group. A designated individual, Personnel C, who will have no involvement in the recruitment or the delivery of interventions, will manage this allocation process. The allocation outcomes will be sealed in envelopes, strictly accessible only to the research team. Trained research personnel A will administer the experimental interventions. Trained research personnel B will administer the control interventions. Trained Research Personnel who administer the interventions will not be blind to the participants' group assignments. Participants will be blinded regarding their group allocation to maintain the study's integrity.

(IV) Data collection:

1. Demographic and past medical history at baseline: Demographic data, including age, sex, education, marital status, religious beliefs and living status, of the patients and their family carers will be collected. Charlson Comorbidity Index will be used to quantify comorbidity, and the Australia-modified Karnofsky Performance Scale will be used to assess the patient's functional ability (Barbetta et al., 2019).
2. The outcomes will be measured using Chinese validated instruments at baseline, 1 and 3 months post-allocation. The repeated-measure design will enable us to examine the short- and long-term intervention effects.

(V) Data Analysis:

1. Quantitative data analysis will be conducted using will be conducted using SPSS 26.0 (IBM, Armonk, NY, USA) for statistical analysis. Descriptive statistical methods will summarise the characteristics of participants and study outcomes. One-way between-group ANOVA will be employed to compare the differences in continuous outcomes between the two study groups. The significance level will be set at 0.05.
2. Qualitative data analysis will be conducted using thematic and content analysis methods. Recordings from qualitative interviews will be transcribed verbatim, coded, and analysed. Qualitative findings will be compared and integrated with the quantitative survey results to provide a more comprehensive research conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years (inclusive) or older.
* Diagnosed with Chronic Obstructive Pulmonary Disease (COPD) by a physician.
* Normal cognitive function.
* Ability to communicate in Mandarin or Cantonese.
* Willingness to participate in the study.

Exclusion Criteria:

* This project will exclude individuals who only partially meet or do not meet the inclusion criteria. Only those who fully meet all inclusion criteria will be invited to participate in the study, and individuals from vulnerable groups or those lacking decision-making capacity will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Patients' decisional conflict regarding EOL care | Before intervention, after intervention and 3-month followup.
  It will be measured using the SURE test to reflect the quality of the decision-making process. This test is derived from the Decisional Conflict Scale. It contains four items that measure uncertainty, inadequate knowledge, unclear values and inadequate support and resources. It is corresponding to the conceptual framework of this study. The response format will be dichotomous (0 = no, 1 = yes), with a higher score indicating a higher level of decisional conflict.

SECONDARY OUTCOMES:
Patients' confidence level regarding three ACP actions - namely, appointing a surrogate and discussing EOL care with a surrogate and medical doctors. | Before intervention, after intervention and 3-month followup.
  Patients' self-efficacy for ACP will be measured using the validated self-efficacy subscale of the ACP Engagement Survey(Liu et al., 2020). This subscale represents one of the four constructs for ACP processes (the other three are knowledge, contemplation and readiness). Participants will rate their confidence level regarding three ACP actions - namely, appointing a surrogate and discussing EOL care with a surrogate and medical doctors - using a five-point Likert scale. A higher score indicates a higher level of self-efficacy.
Patients' readiness for ACP | Before intervention, after intervention and 3-month followup.
  Patients' readiness for ACP will be measured using the validated readiness subscale of the ACP Engagement Survey(Liu et al., 2020). Participants will rate their readiness to complete the ACP as mentioned earlier actions using a five-point scale, from 1 (never thought about it) to 5 (completed already). A higher score indicates a higher level of readiness.
Participant's completion of an Advance Directive (AD) | Before intervention, 3-month followup
  Participant's completion of an Advance Directive (AD) at 3 Months will be determined based on participant self-reports at the 3-month follow-up.
Participants' understanding of the PDA | After intervention and 3-month followup.
  Participants' understanding of the PDA will be measured by asking participants in the experimental group to rate the clarity, linguistic expression, and ease of understanding using a five-point Likert scale. A higher score indicates a higher level of clarity.
Participant's subjective clarity of content, comfort during reading and viewing, and the usefulness of the information of the PDA. | After intervention and 3-month followup.
  Participant's satisfaction with the PDA will be measured by asking participants in the experimental group to rate the clarity of content, comfort during reading and viewing, and the usefulness of the information of the PDA using a five-point Likert scale. A higher score indicates a higher level of satisfaction.
Semi-structured Interviews | After intervention and 3-month followup.
  Participants in the qualitative interview will be recruited by inviting participants from the experimental group using convenience sampling. A trained research personnel will conduct a 30-minute semi-structured interview. The interview will cover topics such as ACP and EOL treatment, concerns regarding medical decision-making, understanding of the ACP process, preferences for various treatment options, and experiences with the PDA. The interviews will adopt experience-sharing methods, allowing participants to express their views, feelings, and experiences freely. All interviews will be voice-recorded and transcribed verbatim for subsequent data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Lai, DN, Principal Investigator — National Taipei University of Nursing and Health Sciences

IPD SHARING:
Plan to Share IPD: No
Data will not be shared to other researchers.

REFERENCES:
- [Background] MacPherson A, Walshe C, O'Donnell V, Vyas A. The views of patients with severe chronic obstructive pulmonary disease on advance care planning: a qualitative study. Palliat Med. 2013 Mar;27(3):265-72. doi: 10.1177/0269216312440606. Epub 2012 Mar 26. PMID 22450158
- [Background] Sapey E, Stockley RA. COPD exacerbations . 2: aetiology. Thorax. 2006 Mar;61(3):250-8. doi: 10.1136/thx.2005.041822. PMID 16517585
- [Background] Momen N, Hadfield P, Kuhn I, Smith E, Barclay S. Discussing an uncertain future: end-of-life care conversations in chronic obstructive pulmonary disease. A systematic literature review and narrative synthesis. Thorax. 2012 Sep;67(9):777-80. doi: 10.1136/thoraxjnl-2012-201835. Epub 2012 Jul 16. PMID 22802331
- [Background] Rietjens JAC, Sudore RL, Connolly M, van Delden JJ, Drickamer MA, Droger M, van der Heide A, Heyland DK, Houttekier D, Janssen DJA, Orsi L, Payne S, Seymour J, Jox RJ, Korfage IJ; European Association for Palliative Care. Definition and recommendations for advance care planning: an international consensus supported by the European Association for Palliative Care. Lancet Oncol. 2017 Sep;18(9):e543-e551. doi: 10.1016/S1470-2045(17)30582-X. PMID 28884703
- [Background] Chan HY, Ng JS, Chan KS, Ko PS, Leung DY, Chan CW, Chan LN, Lee IF, Lee DT. Effects of a nurse-led post-discharge advance care planning programme for community-dwelling patients nearing the end of life and their family members: A randomised controlled trial. Int J Nurs Stud. 2018 Nov;87:26-33. doi: 10.1016/j.ijnurstu.2018.07.008. Epub 2018 Jul 23. PMID 30048916
- [Background] Cheng HB, Shek PK, Man CW, Chan OM, Chan CH, Lai KM, Cheng SC, Fung KS, Lui WK, Lam C, Ng YK, Wong WT, Wong C. Dealing With Death Taboo: Discussion of Do-Not-Resuscitate Directives With Chinese Patients With Noncancer Life-Limiting Illnesses. Am J Hosp Palliat Care. 2019 Sep;36(9):760-766. doi: 10.1177/1049909119828116. Epub 2019 Feb 11. PMID 30744386
- [Background] Bravo G, Trottier L, Arcand M, Boire-Lavigne AM, Blanchette D, Dubois MF, Guay M, Lane J, Hottin P, Bellemare S. Promoting advance care planning among community-based older adults: A randomized controlled trial. Patient Educ Couns. 2016 Nov;99(11):1785-1795. doi: 10.1016/j.pec.2016.05.009. Epub 2016 May 12. PMID 27283764
- [Background] Cohen SM, Volandes AE, Shaffer ML, Hanson LC, Habtemariam D, Mitchell SL. Concordance Between Proxy Level of Care Preference and Advance Directives Among Nursing Home Residents With Advanced Dementia: A Cluster Randomized Clinical Trial. J Pain Symptom Manage. 2019 Jan;57(1):37-46.e1. doi: 10.1016/j.jpainsymman.2018.09.018. Epub 2018 Sep 29. PMID 30273717
- [Background] Michael NG, Georgousopoulou E, Hepworth G, Melia A, Tuohy R, Sulistio M, Kissane D. Patient-caregiver dyads advance care plan value discussions: randomised controlled cancer trial of video decision support tool. BMJ Support Palliat Care. 2022 Jan 25:bmjspcare-2021-003240. doi: 10.1136/bmjspcare-2021-003240. Online ahead of print. PMID 35078875
- [Background] Kim S, Koh S, Park K, Kim J. End-of-life care decisions using a Korean advance directive among cancer patient-caregiver dyads. Palliat Support Care. 2017 Feb;15(1):77-87. doi: 10.1017/S1478951516000808. Epub 2016 Nov 2. PMID 27804916
- [Background] Wen FH, Chen JS, Chou WC, Chang WC, Hsieh CH, Tang ST. Extent and Determinants of Terminally Ill Cancer Patients' Concordance Between Preferred and Received Life-Sustaining Treatment States: An Advance Care Planning Randomized Trial in Taiwan. J Pain Symptom Manage. 2019 Jul;58(1):1-10.e10. doi: 10.1016/j.jpainsymman.2019.04.010. Epub 2019 Apr 18. PMID 31004770
- [Background] Cardona-Morrell M, Benfatti-Olivato G, Jansen J, Turner RM, Fajardo-Pulido D, Hillman K. A systematic review of effectiveness of decision aids to assist older patients at the end of life. Patient Educ Couns. 2017 Mar;100(3):425-435. doi: 10.1016/j.pec.2016.10.007. Epub 2016 Oct 11. PMID 27765378
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics: The Journal of Applied Statistics in the Pharmaceutical Industry. 2005;4(4):287-91.
- [Background] Barbetta C, Allgar V, Maddocks M, Ribeiro C, Wilcock A, Currow DC, Phillips J, Johnson MJ. Australia-modified Karnofsky Performance Scale and physical activity in COPD and lung cancer: an exploratory pooled data analysis. BMJ Support Palliat Care. 2022 Dec;12(e6):e759-e762. doi: 10.1136/bmjspcare-2019-001869. Epub 2019 Jul 11. PMID 31296518
- [Background] Liu L, Zhao YY, Zhang LH, Chan HY. Measuring Self-Efficacy and Readiness for Advance Care Planning in Chinese Older Adults. J Pain Symptom Manage. 2020 Sep;60(3):622-629. doi: 10.1016/j.jpainsymman.2020.06.013. Epub 2020 Jun 20. PMID 32574659